CLINICAL TRIAL: NCT06367153
Title: The Effect of Multiple Doses of BI 1569912 on the Single-dose Pharmacokinetics of Repaglinide, Midazolam and Bupropion Following Oral Administration in Healthy Male and Female Subjects (an Open-label, 2-period Fixed-sequence Trial)
Brief Title: A Study in Healthy Men and Women to Test Whether BI 1569912 Influences the Amount of Repaglinide, Midazolam and Bupropion in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1447-0007; 2023-510461-10-00 (Registry Identifier: CTIS); U1111-1303-9187 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — repaglinide; Midazolam; Bupropion

STUDY DESIGN:
Intervention Model Description: Patients cross over from test treatment (T) to reference treatment (R) (two periods, fixed sequence).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- repaglinide + midazolam + bupropion then BI 1569912 + repaglinide + midazolam + bupropion (Experimental): repaglinide + midazolam + bupropion (reference treatment, R) then BI 1569912 + repaglinide + midazolam + bupropion (test treatment, T)
  Interventions: Drug: BI 1569912; Drug: repaglinide; Drug: midazolam; Drug: bupropion

INTERVENTIONS:
Drug: BI 1569912 — BI 1569912
Drug: repaglinide — repaglinide
Drug: midazolam — midazolam
Drug: bupropion — bupropion

SUMMARY:
The main objective of this trial is to investigate the effect of multiple oral doses of BI 1569912 on the pharmacokinetics of a single oral dose of repaglinide, midazolam and bupropion (i.e. sensitive CYP2C8, CYP3A4 and CYP2B6 substrates).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, standardized mental and neurological assessment, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests without clinically significant abnormalities
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Either male subjects or female subjects who meet the following criteria requiring highly effective contraception from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of adequate contraception, i.e. use of condom (male subjects or male partners of female subjects) plus any of the following methods (female subjects or female partners of male subjects): intrauterine device, hormonal contraception (e.g. implants, injectables, combined oral or vaginal contraceptives), , surgically sterilised (including bilateral tubal occlusion/ligation, hysterectomy, bilateral oophorectomy) or postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of Follicle stimulating hormone (FSH) above 40 U/L is confirmatory)
  * Sexually abstinent (considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments)
  * Vasectomised male subjects or male partners of female subjects (vasectomy at least 1 year prior to enrolment) in combination with a barrier method (i.e. use of condom) and provided that the partner is the sole sexual partner of the trial participant Unprotected sexual intercourse (i.e. without use of condom) of a male subject with a pregnant female partner and sperm donation is not allowed throughout the study and until 30 days after trial completion. Female subjects should not participate in egg donation from the first trial medication administration, for the duration of the study and for at least 30 days after trial completion.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre(s) of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance, in particular hepatic parameters (alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin) or renal parameters (creatinine) exceeding the Upper limit of normal (ULN) after repeated measurements
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke, bulimia or anorexia, or bipolar mood disorder), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 30 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to 30 days
Maximum measured concentration of the analyte in plasma (Cmax) | up to 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com